CLINICAL TRIAL: NCT05939778
Title: A Study on the Efficacy and Safety of Endoscopic Local Injection of Umbilical Cord Mesenchymal Stem Cells（TH-SC01） for the Treatment of Radiation-induced Rectal Injury.
Brief Title: A Study of TH-SC01 in the Treatment of Radiation-induced Rectal Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-SC01-RP-IIT-03
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-09

CONDITIONS: Rectal Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TH-SC01 local injection treatment group (Experimental): The trial was conducted in a non-randomized, single-center, single-arm, dose-escalation design. Three dose groups were preset, which were as follows:
  Low dose group: 3×10^7 live cells/person (6mL); Medium dose group: 6×10^7 live cells/person (12mL) ; High dose group: 1.2×10^8 live cells/person (24mL); Each subject should receive only one corresponding dose. Three subjects were enrolled in the low-dose group,If the safety of the subjects was good, the researchers evaluated the safety and efficacy data and entered the next dose group for treatment. The medium and high-dose groups were enrolled according to the "5+7" principle.
  For the first 3 dose groups, after safety evaluation by the investigators, the maximum dose could reach 2.4×10^8 live cells/person (48mL). If the MTD group is not identified by the highest dose group, it is up to the investigator to decide whether to continue with dose escalation.
  Interventions: Biological: TH-SC01(Umbilical cord mesenchymal stem cells)

INTERVENTIONS:
Biological: TH-SC01(Umbilical cord mesenchymal stem cells) — "5+7" principle:
  1. In medium and high dose groups, 5 subjects were included in each dose group in the first step, and the first 3 subjects had good safety The investigator evaluated safety and efficacy data and could enroll a fourth and fifth subject.
  1. If the number of successful participants in these 5 subjects is less than 2, the study in this dose group will be ended due to drug ineffectiveness, and the researcher will evaluate the safety and enter the next dose group.
  2. If the number of successful participants in these 5 cases is greater than or equal to 2, then proceed to the second step.
  2. 7 subjects were included in the second step.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of allogeneic umbilical cord mesenchymal stem cells in the treatment of radiation-induced rectal injury.

DETAILED DESCRIPTION:
radiation-induced rectal injury (RRI) is a common clinical disease. The symptoms of RRI often include: Abdominal pain, diarrhea, hematochezia, etc., especially chronic radiation-induced late rectal injury (RLRI), are easy to cause the disease to prolong and not heal. Some patients will have severe complications such as massive rectal bleeding, rectal stenosis, intestinal obstruction, deep ulcer, intestinal perforation, and fistula formation after the disease progresses to the advanced stage, most of which occur 2-5 years after the end of radiotherapy. The incidence of radiation rectal injury is high, which has a serious impact on the health and quality of life of patients. Currently, the commonly used treatment methods include non-steroidal anti-inflammatory drugs, mucosal protective agents, hemostatic agents, compound enema preparations, hyperbaric oxygen, surgical treatment, etc., but there is still no standard treatment strategy and effective plan, and clinical treatment is extremely difficult.

Mesenchymal stem cells have the properties of proliferation, differentiation, immune regulation and angiogenesis. There are few clinical studies on the use of mesenchymal stem cells in the treatment of radiation-induced rectal injury. Good therapeutic effect was achieved in vivo and in vitro in the preliminary experiment. The aim of this study was to verify the safety and efficacy of allogeneic mesenchymal stem cells from healthy donors in RRI patients.

Primary objective: To assess the safety (incidence of treatment emergent adverse-events) of TH-SC01.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and sign the informed consent form;
2. Age ≥18 years and <80 years;
3. Patients diagnosed with chronic radiation rectal injury after radiation therapy;
4. Patients with LENT-SOMA scale score ≥1;
5. Good physical condition (WHO functional status score 0-1).

Exclusion Criteria:

1. The patient had severe liver and kidney disease;
2. Severe congestive heart failure or coronary heart disease;
3. Patients have allergic constitutions or severe systemic immune diseases;
4. The patient had active gastrointestinal hemorrhage or acute intestinal obstruction;
5. Patients were pregnant or had other conditions that the investigators deemed unsuitable for inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
lentsoma score scale improved > 0.6 points | 16 weeks
  lentsoma scale can comprehensively reflect the severity of radiation-induced rectal injury from three aspects: subjective feeling, objective situation and intervention measures. There are 14 items in total, each item has a maximum of 4 points, and the final total is divided by 14.

SECONDARY OUTCOMES:
The decreasing level of the Rectal Telangiectasia Density Scale(RTD) | 16 weeks
  The degree of capillary dilatation at the lesion site was observed during colonoscopy. There were four grades, with the highest score being 3.
The declining level of the Vienna Rectoscopy Score | 16 weeks
  The Vienna Rectoscopy Score evaluated the severity of the disease under colonoscopy in five aspects: the degree of telangiectasia, mucosal congestion, ulceration, stenosis, and necrosis. The most serious score is 5 points.
The decreased level ofSemi-quantitative Score of Rectal Radiological Pathological Injury | 16 weeks
  The histological severity of the rectal injury was assessed by colonoscopy. The most severe rating is 10
The decreased levels of SF-36 Scale | 16 weeks
  The quality of life of patients before and after treatment
The decreased levels of Hospital Anxiety and Depression Scales | 16 weeks
  To assess the level of anxiety and depression in the subjects in the hospital
The decreased levels of Visual Analogue Pain Rating Scale | 16 weeks
  The degree of pain is represented by a total of 11 numbers from 0 to 10, 0 means no pain, 10 represents the most pain, according to the degree of pain in the 11 numbers to select a number to represent the pain degree.
Serious adverse event occurred | 2 years
  Cases such as fever, allergy, pain, and severe bleeding should be recorded immediately and treated actively

CONTACTS AND LOCATIONS:
Overall Officials: Fangyu Wang, Study Chair — Director of gastroenterology Department, Jinling Hospital
Locations (1):
- Jinling Hospital, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No